CLINICAL TRIAL: NCT06886724
Title: A Study on the Role of Ligilactobacillus Salivarius LS97 in Modulating Gut Microbiota and Immune System Function
Brief Title: Investigating the Efficacy of Probiotics in Enhancing Gastrointestinal and Immunological Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250307
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Intestinal and Lmmune Function Lmproved
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Intervention with Ligilactobacillus salivarius LS97 (30 billion CFU/day, 3g) was administered daily for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Every day to give 3 g maltodextrin intervention for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial period of this study lasts for 2 months (8 weeks), during which each participant will have 3 visits (at month 0, month 1, and month 2).
  Arms: Probiotic group
Dietary Supplement: Placebo — The trial period of this study lasts for 2 months (8 weeks), during which each participant will have 3 visits (at month 0, month 1, and month 2).
  Arms: Placebo group

SUMMARY:
Evaluate the effectiveness and safety of Ligilactobacillus salivarius LS97 as a food supplement compared to a placebo in improving intestinal and immune functions in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to undergo 3 follow-up visits during the intervention period
2. Be willing to provide blood, urine and stool samples 2 times during the intervention period
3. Good eyesight, can read and write, can wear glasses
4. Have good hearing and be able to hear and understand all instructions during the intervention

Exclusion Criteria:

1. Digestive diseases, mainly gastrointestinal diseases (celiac disease, ulcerative colitis, Crohn's disease)
2. Have a serious neurological condition (epilepsy, stroke, severe head trauma, meningitis in the last 10 years, brain surgery, brain tumor prolonged coma - not including general anaesthesia)
3. Have received/are receiving treatment for the following mental disorders: alcohol/drug/substance abuse dependence, schizophrenia psychosis, bipolar disorder
4. Take medication for depression or low mood
5. Internal organ failure (heart, liver or kidney failure, etc.)
6. Have received radiation or chemotherapy in the past
7. have undergone a general anesthesia procedure/procedure within the past three years, or plan to undergo a general anesthesia procedure/procedure within the next 3 months during this trial period
8. Have had hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the composition of fecal microbiota before and after intervention. | Week 0 and Week 8
  Analyzed by 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Xu fei, Zhengzhou, Henan, China